CLINICAL TRIAL: NCT07081568
Title: Research on Binaural Synchronous Vagus Nerve Regulation of Sensorimotor Disorders After Cerebral Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchang University Affiliated Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Wentao Zeng, Doctor of Medicine, Nanchang University Affiliated Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFYLL-KY-PJ-2025-004
Record Dates: First submitted 2025-06-19; First posted 2025-07-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Infarction
Keywords: Ischemic Stroke; Transcutaneous Auriculai Vagus Nerve Stimulation; Rehabilitation for Cerebral Infarction; Neuromodulation
MeSH Terms: conditions — Cerebral Infarction; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Stimulation Group (No Intervention): Sham Stimulation Group received sham stimulation using device B, which had identical appearance, interface parameters, and physical sensation but no therapeutic effect. Stimulation parameters were set as follows: sinusoidal waveform; pulse width of 200μs; frequency of 20Hz; current adjusted to 0mA by the investigator; single session duration of 30 minutes. After each session, the device was disinfected with 75% alcohol. Treatment was administered once daily, 5 days per week, for a total duration of 4 weeks.
- transcutaneous auriculai vagus nerve stimulation (Experimental): The patient was positioned in a supine position. Two stimulating electrodes were placed on the bilateral concha cymba and concha cavum. Stimulation parameters were set as follows: sinusoidal waveform; pulse width of 200μs; frequency of 20Hz; initial intensity of 2mA. Each treatment session lasted 30 minutes. Treatment was administered once daily, 5 days per week, for a total duration of 4 weeks. After each treatment session, the device was disinfected with 75% alcohol.
  Interventions: Device: transcutaneous auriculai vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auriculai vagus nerve stimulation — During bi-ear synchronous vagus nerve stimulation, the patient was positioned in a supine position. Two stimulating electrodes were placed bilaterally in the concha cymba and concha cavum of the ears. The patient received treatment for 30 minutes per session, once daily, 5 days per week, for a total of 4 weeks. Following each treatment session, the device was disinfected with 75% alcohol.
  Arms: transcutaneous auriculai vagus nerve stimulation

SUMMARY:
The aim of this study is to determine the efficacy and safety of binaural synchronous vagus nerve regulation in the treatment of patients with sensory and motor dysfunction after cerebral infarction through a randomized controlled clinical study, and to provide high-quality evidence support for binaural synchronous vagus nerve regulation in the treatment of cerebral infarction.

DETAILED DESCRIPTION:
The research subjects were first-onset cerebral infarction and were recruited at the Affiliated Rehabilitation Hospital of Nanchang University (the Fourth Affiliated Hospital). Based on the estimated sample size, a total of 40 patients were included in this study. The randomization grouping protocol divided 40 patients into the experimental group and the control group in a 1:1 ratio. Experimental group: Received synchronous vagus nerve regulation in both ears. Control group: Received false stimulation. The randomization procedure was carried out by independent statisticians who were not involved in the implementation and statistics of the study. The trial secretary placed the generated random numbers and groups respectively into opaque envelopes. After the patients were confirmed to be included in the group, the project leader opened the envelopes numbered in sequence to complete the grouping. This study was A double-blind design, using a unified binaural vagus nerve electrical stimulation device (JY-VNS-200, Jiangxi Jingyi Medical Technology Company Limited.). To achieve researcher blindness, the device was preset in A/B mode, with one mode being true stimulation and the other mode being false stimulation. After the experiment, unblinding was performed by personnel who were not involved in the study. During the experiment, the patients did not know whether they were receiving actual treatment or a placebo. The patients were blind. Meanwhile, the evaluators and statistical analysts were unaware of the grouping of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first-episode ischemic stroke within 7 to 14 days of onset;
* Be over 18 years old;
* The skin at the irritated area remains intact;
* The informed consent form has been signed.

Exclusion Criteria:

* Severe cognitive dysfunction (Mini-Mental State Examination≥19);
* Peripheral limb movement limiting factors (fractures);
* History of major neurological and mental disorders in the past;
* Uncontrollable limb and facial muscle twitching, and spontaneous profuse sweating;
* Intracranial shunt pumps, metal implants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor function score | Before the start of treatment, the last week before the end of treatment, and the third month after the onset of the disease
  Motor function was evaluated using the Fugl-Meyer Assessment of Motor Recovery after Stroke (FMA) .The assessment was performed three times. The minimum score for the Fugl-Meyer Assessment (FMA) is 0, and the maximum score is 226.A higher score on the FMA indicates better motor recovery/function and a lower level of motor impairment.
Overall functional score | Before the start of treatment, the last week before the end of treatment, and the third month after the onset of the disease
  Assess three times using the National Institutes of Health Stroke Scale. The maximum score on the scale is 42, and the minimum score is 0.Higher scores denote more severe stroke symptoms.
Transcranial Magnetic Stimulation combined with Electroencephalography（TMS-EEG） | Before the start of treatment, the last week before the end of treatment, and the third month after the onset of the disease
  Amplitude and latency of key TMS-evoked potential (TEP) components ( N100, P180, N200) recorded from specific scalp electrodes (Fz, Cz, Pz) following single-pulse TMS over the dorsolateral prefrontal cortex (DLPFC).
Sensory function score | Before the start of treatment, the last week before the end of treatment, and the third month after the onset of the disease
  Using the Eastern Michigan Neuropathy Symptom Score Assessment sensory scale for assessment, the lowest possible score is 0 and the highest is 100. A higher score indicates that the patient's neurological symptoms are more severe and that the degree of nerve damage is more apparent.

SECONDARY OUTCOMES:
Cognitive function score | Before the start of treatment
  Using the Mini-Mental State Examination scale for assessment, the minimum score is 0 and the maximum score is 30. The higher the score, the better the cognitive function of the examinee, indicating a normal cognitive state.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Rehabilitation Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No